CLINICAL TRIAL: NCT01938352
Title: Randomised, Double-Blind, Placebo-Controlled, Phase IIa Study in Healthy Volunteers to Evaluate the Protective Efficacy and Safety of CR8020 in an Influenza Challenge Model
Brief Title: Evaluation of the Protective Efficacy and Safety of CR8020 in an Influenza Challenge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Collaborators: Retroscreen Virology Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR102595; CRU-CS-001; CR8020FLZ2002 (Other: Crucell Holland BV); 2013-002185-39 (EudraCT Number)
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-03

CONDITIONS: Influenza
Keywords: Influenza; Virus; Monoclonal Antibody; Immunization; Treatment
MeSH Terms: conditions — Influenza, Human; Virus Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- CR8020 (Experimental): CR8020 administered as a single 2-hour intravenous infusion
  Interventions: Biological: CR8020
- Placebo (Placebo Comparator): Placebo administered as a single 2-hour intravenous infusion
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CR8020 — CR8020 15 mg/kg, administered by intravenous infusion
  Arms: CR8020
Biological: Placebo — Placebo (hydrous dextrose in water for injection), administered by intravenous infusion
  Arms: Placebo

SUMMARY:
After prophylactic vaccination with CR8020, a monoclonal antibody, subjects will be challenged with the H3N2 virus. The protective efficacy, safety, tolerability, pharmacokinetics, and potential immunogenicity will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ≥ 18 and ≤ 45 years of age.
2. In good health, with no major medical conditions from medical history, physical examination, and routine laboratory tests as determined by the Investigator at a screening evaluation.
3. A total body weight ≥50 kg and a BMI of >18. If the BMI is above 28 the subject may be included if the waist measurement is less than 94 cm (male), or less than 80 cm (female).
4. (a) Male subjects must use highly effective contraception consisting of two forms of birth control (one of which must be a barrier method) starting at entry to Quarantine until after the Day 96 (± 5 days) Follow-up Visit.

   (b) In addition, male subjects must not donate sperm following discharge from Quarantine until after the Day 96 (± 5 days) Follow-up Visit.

   (c) Female subjects must be either:
   * Documented status as surgically sterile or post hysterectomy or-
   * If of childbearing potential, must have a negative serum and urine pregnancy test at study specific screening and Day -4/-3 and must be using highly effective contraception consisting of two forms of birth control (one of which must be a barrier method) starting at entry to Quarantine and continue until the Day 96 (± 5 days) Follow-up Visit.

   Acceptable forms of effective contraception include:
   * Established use of oral, injected or implanted hormonal methods of contraception
   * Placement of an intrauterine device (IUD) or intrauterine system (IUS).
   * Barrier methods of contraception: Condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
   * Male sterilisation (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). [For female subjects on the study, the vasectomised male partner should be the sole partner for that subject].

   True abstinence: When this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception].
5. An informed consent document signed and dated by the subject and Investigator.
6. Sero-suitable for challenge virus.

Exclusion Criteria:

1. Subjects who have a significant history of tobacco use at any time (≥ total 10 pack year history, e.g. one pack a day for 10 years)
2. (a) Females who are pregnant or have been pregnant within six months prior to the study, or who have been breastfeeding within three months prior to screening. Females who have a positive pregnancy test at any point in the study will be withdrawn immediately.

   (b) Females intending to become pregnant within three months of administration of CR8020 or placebo or males with female partners intending to become pregnant within three months of administration of CR8020 or placebo
3. Any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinological, haematological, hepatic, immunological, metabolic, urological, neurological, psychiatric, renal, and/or other major disease or malignancy, as judged by the Investigator

   1. Eczema/Atopic Dermatitis: (Subjects with clinically mild eczema/atopic dermatitis may be included at the Investigator's discretion e.g. if there is no regular use of topical steroids, no eczema in cubital fossa)
   2. Psoriasis:(Subjects with active psoriasis affecting less than 5% of the body's surface area for the past five years can be included at the Investigator's discretion- (1% of the body area is roughly equivalent to the palm of the subject's hand). Patients with a history of completely resolved guttate psoriasis can be included)
   3. Psychiatric: (Subjects with a diagnosis of a single mild or moderate depressive episode two or more years ago, with good evidence of preceding stressors and which resolved within approximately three months (i.e. reactive depression), may be included at the Investigator's discretion)
4. Abnormal pulmonary function in the opinion of the Investigator as evidenced by clinically significant abnormalities on spirometry
5. History or evidence of autoimmune disease or known immunodeficiency of any cause
6. Subjects with any history of asthma, chronic obstructive pulmonary disease (COPD), pulmonary hypertension, reactive airway disease, or chronic lung condition of any aetiology (See No. 7 for asthma)
7. Asthma (A history of childhood asthma before the age of 12 is acceptable provided the subject is asymptomatic without treatment. Patients with a single episode of wheezing after age 12 (lasting less than eight weeks) can be included at the Investigator's discretion)
8. Positive human immunodeficiency virus (HIV), Hepatitis A (HAV), B (HBV), or C (HCV) test
9. Any significant abnormality altering the anatomy of the nose or nasopharynx
10. Any clinically significant history of epistaxis
11. Any nasal or sinus surgery within six months of Viral Challenge
12. Recurrent history of clinically significant autonomic dysfunction
13. Any abnormal laboratory test or ECG which is deemed by the Investigator to be clinically significant
14. Confirmed positive test for drugs of abuse deemed by the Investigator to be clinically significant
15. Venous access deemed inadequate for the phlebotomy and cannulation demands of the study
16. Known allergy to any of the following:

    * excipients in the Challenge Virus inoculum
    * any CR8020 excipients (sucrose, L-histidine L-histidine monohydrochloride, polysorbate 20)
    * oseltamivir or other influenza treatments
17. Health care workers (e.g. doctors, nurses, medical students and allied healthcare professionals) who work in units with severely immuno-compromised patients (e.g. bone marrow transplant units)
18. Presence of household member or close contact(s) (for an additional two weeks after discharge from the isolation facility) who:

    * has known immunodeficiency
    * is receiving immunosuppressant medication
    * is undergoing or soon to undergo cancer chemotherapy within 28 days of Viral Challenge
    * has been diagnosed with emphysema, COPD, or other severe lung disease and resides in a nursing home
    * has received a bone marrow or solid organ transplant
19. Evidence of vaccinations within the four weeks prior to Human Viral Challenge. Intention to receive travel vaccination(s) before the Day 96 (± 5 days) Follow Up Visit
20. Those employed or immediate relatives of those employed at Retroscreen Virology Limited or the Sponsor
21. Receipt of blood or blood products, or loss (including blood donations) of 450 mL or more of blood, during the three months prior to Viral Challenge or planned donation/receipt throughout the course of the study
22. Use of nasal steroids within 28 days prior to Viral Challenge Use of any other medication or product (prescription or over-the-counter), for symptoms of hay fever, rhinitis, nasal congestion or respiratory tract infection within seven days of Viral Challenge
23. Receipt of any investigational drug within three months prior to Viral Challenge Prior participation in a clinical trial with the same strain of respiratory virus Participation in any other Human Viral Challenge study with a respiratory virus within one year prior to the day of Viral Challenge
24. Receipt of systemic glucocorticoids, antiviral drugs, or immunoglobulins (Igs) or any other cytotoxic or immunosuppressive drug within six months prior to dosing, or receipt or any systemic chemotherapeutic agent at any time
25. Previous receipt of monoclonal antibodies or monoclonal antibody fragments at any time
26. Presence of significant respiratory symptoms existing on the day of challenge or between admission to the unit and inoculation with the Challenge Virus History suggestive of respiratory infection within 14 days prior to admission to the Quarantine Unit
27. Any other finding that, in the opinion of the Investigator or Sponsor, deems the subject unsuitable for the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2013-10-02 (Actual); Primary Completion 2014-01-22 (Actual); Study Completion 2014-01-22 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of viral load | Day 7
  Measured from the nasopharyngeal mucosa (by qPCR) post influenza virus challenge

CONTACTS AND LOCATIONS:
Locations (1):
- London, United Kingdom